CLINICAL TRIAL: NCT06182631
Title: A Randomized Clinical Trial of Buzzy Versus Vapocoolant in Pain Relief During Phlebotomy and IV Catheterization in the Pediatric ED
Brief Title: Clinical Trial Testing Buzzy Bee vs Vapocoolant During IV Placement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jill C Fennell, Pediatric Emergency Medicine Fellow, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00002993
Record Dates: First submitted 2023-04-18; First posted 2023-12-27 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Intravenous Administration
Keywords: analgesic; anxiolytic; Buzzy Bee; Shot-blocker

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Vapocoolant (Experimental): Will have nurse spray vapocoolant on the skin before IV insertion, will then videotape patient and ask them and parent to fill out FACES form.
  Interventions: Drug: Vapocoolent
- Buzzy Bee (Experimental): Will have nurse put Buzzy Bee on arm before, and leave it on during IV insertion. Will then videotape patient and ask them and parent to fill out FACES form.
  Interventions: Device: Buzzy Bee
- Placebo (Placebo Comparator): Will have nurse place a rubber band around arm before IV insertion. Will then videotape patient and ask them and parent to fill out FACES form.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Buzzy Bee — The Buzzy is a vibrating palm-sized device with removable ice wings developed by MMJ Labs Atlanta, GA. It uses Melzack and Wall's Gait Control theorywhich asserts that activation of non-nociceptive fibers can interfere with signals from pain fibers thereby inhibiting pain.
  Arms: Buzzy Bee
Drug: Vapocoolent — Vapocoolent is a volatile refrigerated liquid, ie ethyl chloride, which is supposed to feel like the skin is numb before insertion of the IV.
  Arms: Vapocoolant
Other: Placebo — A band will be placed on the arm before IV insertion for placebo effect.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the anxiety and pain levels of patients when using Buzzy with ice, Vapocoolant, and placebo when inserting IV's line for IV fluids and/or phlebotomy in pediatric patients in the pediatric emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Need IV's line placement for IV fluids and/or phlebotomy

Exclusion Criteria:

* patients sensitive to cold i.e. Raynaud's
* critically ill patients
* mentally challenged patients
* GCS< 15
* Patient with altered sensation
* Patients needing more than one attempt at IV placement

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 172 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oshei Childrens Hospital, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bijttebier P, Vertommen H. The Impact of Previous Experience on Children's Reactions to Venepunctures. J Health Psychol. 1998 Jan;3(1):39-46. doi: 10.1177/135910539800300103. PMID 22021341
- [Background] Blount R. L., Zempsky W. T., Jaaniste T., Evans S., Cohen L. L., Devine K. A., Zeltzer L. K. Management of pain and distress due to medical procedures. In: Roberts M C, Steele R, editors. Handbook of pediatric psychology. 4th Ed. New York: Guilford Press; 2009. pp. 171-188.
- [Background] Cohen Reis E, Holubkov R. Vapocoolant spray is equally effective as EMLA cream in reducing immunization pain in school-aged children. Pediatrics. 1997 Dec;100(6):E5. doi: 10.1542/peds.100.6.e5. PMID 9374583
- [Background] Hamilton JG. Needle phobia: a neglected diagnosis. J Fam Pract. 1995 Aug;41(2):169-75. PMID 7636457
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Lunoe MM, Drendel AL, Levas MN, Weisman SJ, Dasgupta M, Hoffmann RG, Brousseau DC. A Randomized Clinical Trial of Jet-Injected Lidocaine to Reduce Venipuncture Pain for Young Children. Ann Emerg Med. 2015 Nov;66(5):466-74. doi: 10.1016/j.annemergmed.2015.04.003. Epub 2015 Apr 29. PMID 25935844
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Pate J.T., Blount R.L., Cohen L.L. & Smith A.J. (1996). Childhood medical experience and temperament as predictors of adult functioning in medical situations. Child Health Care, 25 (4): 281-298.
- [Background] Shah V, Taddio A, Rieder MJ; HELPinKIDS Team. Effectiveness and tolerability of pharmacologic and combined interventions for reducing injection pain during routine childhood immunizations: systematic review and meta-analyses. Clin Ther. 2009;31 Suppl 2:S104-51. doi: 10.1016/j.clinthera.2009.08.001. PMID 19781433

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 221 Patients were approached by research assistants in the Emergency Department, 37 refused consent and 5 excluded due to medical reasons
Pre-assignment Details: 7 patients were then excluded due to multiple IV attempts
Period: Overall Study
Arm/Group | Vapocoolant | Buzzy Bee | Placebo
Started | 57 | 56 | 58
Completed | 57 | 56 | 58
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vapocoolant | Buzzy Bee | Placebo | Total
Number analyzed (Participants) | 57 | 56 | 58 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 57 | 56 | 58 | 171
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (4.1) | 12.6 (3.8) | 12.7 (4) | 12.6 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 27 | 38 | 98
  Male | 24 | 29 | 20 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 11 | 5 | 23
  White | 45 | 37 | 49 | 131
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 57 | 56 | 58 | 171

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Based on Wong-Baker Pain Scale During IV Placement With Buzzy Bee or Vapocoolent
Description: Wong- Baker Faces Pain Scale with scores: scale is 0-10, with 0 being no pain and 10 maximum pain. The changes in pain between the treatment groups were analyzed using chi square and one-way ANOVA for categorical and continuous variables respectively. Pre and post FACES pain scale-revised were reported as means and standard deviations
Time Frame: post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Vapocoolant: use of vapocoolant for IV placement
- Buzzy Bee: Use of Buzzy Bee for IV placement
- Placebo: IV placement without use of buzzy bee or vapocoolant
Arm/Group | Vapocoolant | Buzzy Bee | Placebo
Number analyzed (Participants) | 57 | 56 | 58
units on a scale
  Pre-intervention | 4.54 (2.65) | 5.41 (2.9) | 5.03 (3.01)
  Post-intervention | 3.84 (3.12) | 3.58 (2.87) | 4.57 (3.43)

2. Primary Outcome: Perceived FACES Pain Score in Sensation of Pain During IV by Parent or Care-giver
Description: Faces Pain Scale revised with scores: scale is 0-10, with 0 being no pain and 10 maximum pain.
Time Frame: post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vapocoolant | Buzzy Bee | Placebo
Number analyzed (Participants) | 57 | 56 | 58
units on a scale
  Pre-intervention | 3.06 (2.98) | 3.46 (2.88) | 2.86 (2.85)
  Post-intervention | 2.24 (2.56) | 1.69 (2.28) | 2.79 (2.84)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during patient stay, an average of 3 hours
Arm/Group | Vapocoolant | Buzzy Bee | Placebo
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56 | 0/58
Other Adverse Events (participants affected / at risk) | 0/57 | 0/56 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT06182631/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT06182631/ICF_001.pdf